CLINICAL TRIAL: NCT03752840
Title: Village-Integrated Eye Worker Trial II (VIEW II):A Cluster-randomized Trial of the Effectiveness of Community-based Ocular Disease Screening
Brief Title: Village-Integrated Eye Worker Trial II
Acronym: VIEW II
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Seva Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 17-22776-2
Record Dates: First submitted 2018-11-16; First posted 2018-11-26 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Age-related Macular Degeneration; Diabetic Retinopathy; Glaucoma
MeSH Terms: conditions — Macular Degeneration; Diabetic Retinopathy; Glaucoma | interventions — Visual Acuity; Tomography, Optical Coherence; Intraocular Pressure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Screening (Experimental)
  Interventions: Other: Visual acuity (presenting and pinhole); Other: Optical coherence tomography (OCT); Other: Intraocular pressure; Other: Active linkage to care; Other: Fundus Photography
- Case detection (Active Comparator)
  Interventions: Other: Visual acuity (presenting and pinhole)

INTERVENTIONS:
Other: Visual acuity (presenting and pinhole) — Presenting and pinhole visual acuity will be assessed using the Peek Acuity mobile application. Participants meeting referral criteria will be referred to the nearest eye care center or eye hospital.
Other: Optical coherence tomography (OCT) — OCT will be used to image the anterior segment, the macula, and the retinal nerve fiber layer. The images will be assessed for abnormalities and participants meeting referral criteria will be referred to the local eye hospital.
  Arms: Screening
Other: Intraocular pressure — Intraocular pressure will be measured using an iCare tonometer. Participants meeting referral criteria will be referred to the nearest eye care center or eye hospital.
  Arms: Screening
Other: Active linkage to care — Referred participants will be followed closely by study staff to ensure completion of follow-up visits.
  Arms: Screening
Other: Fundus Photography — Fundus cameras will be used to image the macula and optic nerve. The images will be assessed for abnormalities and participants meeting referral criteria will be referred to the local eye hospital.
  Arms: Screening

SUMMARY:
The vast majority of blindness is avoidable. The World Health Organization (WHO) estimates that 80% of cases of visual impairment could be prevented or reversed with early diagnosis and treatment. The leading causes of visual impairment are cataract and refractive error, followed by glaucoma, age-related macular degeneration (AMD), and diabetic retinopathy (DR). Loss of vision from these conditions is not inevitable; however, identifying cases early and linking cases with appropriate care remain significant challenges.

To address the global burden of avoidable blindness, eye care systems must determine optimal strategies for identifying people with or predisposed to visual impairment beyond opportunistic screening. Outreach programs can prevent blindness both by screening for asymptomatic disease like age-related macular degeneration (AMD), diabetic retinopathy (DR), and glaucoma and case detection of symptomatic disease like cataract and refractive error. Eye care systems have developed numerous approaches to these identification methods, including screening using telemedicine and case detection via cataract camps or health worker models, but no studies have been conducted on the comparative effectiveness or cost effectiveness of these various approaches.

Technology promises to greatly improve access to sophisticated eye care. AMD, DR, and glaucoma can result in irreversible vision loss, and early diagnosis and effective treatment can prevent progression. Thus, mass screening programs may prevent progression and improve the vision of a population. However, mass screening for eye disease is currently not recommended. Although self-evident that early detection can prevent blindness for an individual, no randomized controlled trial has been able to demonstrate that screening improves visual acuity at the regional level. However, recent technological advances promise to dramatically change the equation by allowing non-medical personnel to use mobile, easy-to-use retinal imaging devices to diagnose screenable eye diseases such as AMD, DR, and glaucoma. Mobile technology could also transform the way clinics communicate with their patients, improving linkage to and retention in care.

Optical coherence tomography (OCT) is an ideal test for screening. OCT can be performed through an undilated pupil and is less subject to optical aberrations due to cataract than is fundus photography. OCT machines have pre-installed algorithms to screen for glaucoma, and major anatomical abnormalities can easily be detected even by novice technicians. The infrared image allows detection of referable diabetic retinopathy, and newer OCT angiography machines offer even more discrimination of early diabetic retinopathy. OCT machines are ever more portable, and could be feasibly used in mobile screening programs.

The investigators propose a large cluster-randomized trial to compare two population level blindness prevention programs: (1) a state-of-the-art screening program employing OCT, fundus photography, and intraocular pressure testing to screen for glaucoma, DR, and AMD followed by enhanced linkage-to-care to the local eye hospital, and (2) a screening program involving only visual acuity assessment. An initial door-to-door census will assess baseline visual acuity in both study arms. The investigators will compare visual acuity between the two arms through a second door-to-door census 9 years later (primary outcome).

DETAILED DESCRIPTION:
The research will consist of a large cluster-randomized trial in which all clusters receive visual acuity screening during a baseline census, and then half subsequently receive screening with OCT, fundus photography, and intraocular pressure testing with an iCare tonometer. Participants with abnormal results will be referred to the local eye hospital for examination and treatment. Repeat visual acuity assessment will be performed 9 years later. Those with visual impairment at the time of the final census, defined as visual acuity worse than Snellen 20/60 (Metric Snellen worse than 6/18; logMAR worse than 0.48), will receive a comprehensive eye exam to determine the cause of visual impairment.

Specific Aim 1 - Visual Acuity: To determine whether an intensive screening program results in better visual acuity at 9 years than screening with visual acuity testing alone. The investigators hypothesize that individuals from clusters randomized to the intensive screening program will have better visual acuity compared to those receiving visual acuity testing alone.

Specific Aim 2 - Eye Disease: To determine whether an intensive screening program reduces the incidence of visual impairment due to AMD, DR, or glaucoma. The investigators hypothesize that incident visual impairment due to AMD, DR, or glaucoma will be less common in clusters randomized to the intensive screening program.

ELIGIBILITY:
Community level

Inclusion Criteria:

* Located in catchment area of Bharatpur Eye Hospital or Lumbini Eye Institute
* Reachable by non-4WD vehicle
* Urban or peri-urban

Exclusion Criteria:

- Local leaders unwilling to participate

Person level

Inclusion Criteria:

* 50 years and older
* Residing in the community during the time of the census

Exclusion Criteria:

- Unwilling to participate

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60200 (Estimated)
Dates: Start 2019-04-21 (Actual); Primary Completion 2029-08-31 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
Pinhole visual acuity (logMAR) in people aged 50 years and older | 9 years
  Visual acuity will be assessed using the Peek Acuity mobile application during the final census.

SECONDARY OUTCOMES:
Incidence of visual impairment due to AMD, DR, or glaucoma | 9 years
  Participants with incident visual impairment, defined as Snellen worse than 20/60 (Metric Snellen worse than 6/18; logMAR worse than 0.48), at the time of the final census will receive a comprehensive eye exam to determine the cause of visual impairment
Bilateral blindness in people aged 50 years and older, defined as pinhole visual acuity worse than Snellen 20/400 (Metric Snellen worse than 6/120; logMAR worse than 1.3) in the better-seeing eye | 9 years
  Visual acuity will be assessed using the Peek Acuity mobile application during the final census.
Presenting visual acuity (logMAR) in people aged 50 years and older | 9 years
  Visual acuity will be assessed using the Peek Acuity mobile application during the final census.
Cost-effectiveness of the screening intervention | 9 years
  Costs associated with the screening intervention will be actively recorded during the study period and number of cases of AMD, DR, and glaucoma diagnosed and visual acuity as assessed with Peek Acuity during the final census will be used to evaluate effectiveness.

OTHER OUTCOMES:
Bilateral visual impairment in people aged 50 years and older, defined as pinhole visual acuity worse than Snellen 20/60 (Metric Snellen worse than 6/18; logMAR worse than 0.48) in the better-seeing eye | 9 years
  Visual acuity will be assessed using the Peek Acuity mobile application during the final census.
Bilateral presenting visual impairment in people aged 50 years and older, defined as presenting visual acuity worse than Snellen 20/60 (Metric Snellen worse than 6/18; logMAR worse than 0.48) in the better-seeing eye | 9 years
  Visual acuity will be assessed using the Peek Acuity mobile application during the final census.
Bilateral presenting blindness in people aged 50 years and older, defined as presenting visual acuity worse than Snellen 20/400 (Metric Snellen worse than 6/120; logMAR worse than 1.3) in the better-seeing eye | 9 years
  Visual acuity will be assessed using the Peek Acuity mobile application during the final census.

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Keenan, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared with other investigators upon request after the conclusion of the study. A request form will be available on Open Science Framework (https://osf.io/fgvrt/); all requests will be approved by the executive committee of the trial before sharing data. GPS data will not be shared.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: De-identified data will be shared after publication of the major findings of the study, which we anticipate will occur around 6 months after the study conclusion.
Access Criteria: De-identified data will be available upon request.
URL: https://osf.io/fgvrt/

REFERENCES:
- [Derived] O'Brien KS, Stevens VM, Byanju R, Kandel RP, Bhandari G, Bhandari S, Melo JS, Porco TC, Lietman TM, Keenan JD; Group Information for the VIEW II Study Group. Cluster-randomised trial of community-based screening for eye disease in adults in Nepal: the Village-Integrated Eye Worker Trial II (VIEW II) trial protocol. BMJ Open. 2020 Oct 15;10(10):e040219. doi: 10.1136/bmjopen-2020-040219. PMID 33060092